CLINICAL TRIAL: NCT01315951
Title: Petrolatum's Effect on Initial Symptoms of Nonscalp Seborrheic Dermatitis and Preventing Exacerbation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Ryan D Stevenson left Organization (Genesys) prior to Ascension acquiring record; no evidence of completion
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Jackie Kirchen, Director research integrity and compliance, Ascension Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME 10 0054
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Seborrheic Dermatitis
Keywords: Non scalp Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — Petrolatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Petroleum Jelly (Experimental): Every patient will be applying petroleum jelly to the affected areas per protocol.
  Interventions: Biological: Petroleum Jelly

INTERVENTIONS:
Biological: Petroleum Jelly — Every patient will be instructed to wet the affected area, blot dry, and then apply petroleum jelly to the area before bedtime. This regimen is to be followed every other night until symptoms diminish. The patient should follow-up at one week, two weeks, and four weeks after treatment begins to see the outcome.
  Other Names: Petrolatum, Vaseline

SUMMARY:
The goal of this research is to demonstrate the use of petroleum jelly in prevention of nonscalp seborrheic dermatitis exacerbations at the first signs of a flare. In doing so, it will decrease the chronic use of topical steroids. The use of petrolatum should have favorable outcomes for patients, without the side-effects.

DETAILED DESCRIPTION:
Nonscalp seborrheic dermatitis (NSSD) is typically a benign inflammatory process of the skin that affects oil rich areas including in and between eyebrows, paranasal area, behind ears, over the sternum, and groin. While these lesions typically come and go without proposing a threat to the patient, they can be socially debilitating, and psychologically distressing.

The mainstay treatment for an exacerbation of NSSD is topical steroids. Topical steroids are very effective and useful to patient's who are desperately seeking treatment. However, most family practitioners are reluctant to prescribe or recommend topical steroids for chronic conditions like NSSD due to the potential side-effects including permanent atrophy of the skin.

NSSD has an unknown etiology. However, one of its biggest risk factors appears to be dry skin due to its increase in incidence during colder seasons, and with use of alcohol-containing topicals. Naturally occurring skin yeast (ie Malassezia) are also thought to play a part.

Petrolatum is considered a skin protectant and has a strong ability to hold moisture in skin. Along with restricting water from leaving skin, it also decreases most air from contacting the skin. This may slow the growth and activity of skin yeast that are typically considered facultative anaerobes.

A patient diagnosed with nonscalp seborrheic dermatitis will be consented into the study and given instructions on the petroleum treatment. This includes wetting the affected area, blotting dry, and then applying petrolatum to the area before bedtime. This regimen is to be followed every other night until symptoms diminish. The patient will come back to the office for follow-up at one week, two weeks, and four weeks after treatment begins to see the outcome. Pictures will be taken at each encounter and used to measure progress through one mm graphs. Patients will not be identifiable in these pictures, and they will be labeled with the patient's given ID number.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old who are patients of the Genesys East Flint Clinic and have been diagnosed with recurrent NSSD
* Patients are to use the petrolatum treatment strictly for the initial symptoms of NSSD: Excessive flaking, and erythematous macules or papules
* Patients who are able to attend the follow-up appointments for assessment
* Patients are to have the doctor's confidence that that patient will correctly implement the treatment plan

Exclusion Criteria:

* Patients not in the 18-75 years of age range.
* Patients who are receiving treatment for their seborrheic dermatitis (Scalp or nonscalp) elsewhere.
* Patients who have not demonstrated recurrent NSSD.
* Patients who are unable to commit to a follow-up appointments for assessment.
* Patients who do not have the physician's confidence in implementing the studies treatment plan effectively.
* Patient's who are unable/unwilling to have petrolatum on affected area for at least a 6 hour length of time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Measuring the Effectiveness of Petroleum Jelly in Treating Nonscalp Seborrheic Dermatitis | 4 weeks
  Petroleum jelly will be applied to the areas of the face affected by Nonscalp Seborrheic Dermatitis every other night for four weeks. Patients will be seen in the office at one week, two weeks, and one month during the course of the treatment. Pictures will be taken at each visit to determine the progress of the treatment.

SECONDARY OUTCOMES:
Patient Satisfaction ofTreatment | 4 weeks
  Patients will be surveyed initially when they are consented asking about their personal history of nonscalp seborrheic dermatitis including triggers and previous and current treatment measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D Stevenson, BS, Principal Investigator — Ascension Health
Locations (1):
- Genesys East Flint Campus, Burton, Michigan, United States